CLINICAL TRIAL: NCT05161481
Title: Randomised, Double-blind, Placebo-controlled and Parallel Group Trial to Investigate the Effects of Two Doses (Up-titration to a Fixed Dose Regimen) of Oral BI 685509 on Portal Hypertension After 24 Weeks Treatment in Patients With Clinically Significant Portal Hypertension (CSPH) in Compensated Cirrhosis
Brief Title: A Study to Test Whether Two Different Doses of Avenciguat Help People With Liver Cirrhosis and High Blood Pressure in the Portal Vein (Main Vessel Going to the Liver)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1366-0021; 2021-001285-38 (EudraCT Number)
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hypertension, Portal
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Avenciguat 2 mg BID (Experimental): Participants received Avenciguat combined with matching placebo tablets twice daily (BID). At Visit 2 (Week 1), each dose included one 1 mg Avenciguat tablet and one 2 mg placebo tablet (four tablets daily). At Visit 3 (Week 2), the dose was up titrated to 2 mg Avenciguat BID (one 1 mg placebo tablet and one 2 mg Avenciguat tablet (four tablets daily)). From Visit 4 onward (Week 3+), a pseudo up-titration was applied, with participants taking one 2 mg Avenciguat tablet and one 3 mg placebo tablet per dose (four tablets daily) to maintain blinding. This regimen continued for 24 weeks, with doses taken with water, with or without food.
  Interventions: Drug: Avenciguat (BI 685509)
- Avenciguat 3 mg BID (Experimental): Participants received Avenciguat with matching placebo tablets twice daily (BID). At Visit 2 (Week 1), each dose contained one 1 mg Avenciguat tablet and one 2 mg placebo tablet (four tablets daily). At Visit 3 (Week 2), the dose was up titrated to 2 mg Avenciguat BID (one 1 mg placebo tablet and one 2 mg active tablet (four tablets daily)). From Visit 4 onward (Week 3+), the dose was further up titrated to 3 mg Avenciguat BID (one 2 mg placebo tablet and one 3 mg active tablet per dose (four tablets daily)). This regimen was maintained for 24 weeks, with doses taken with water, with or without food.
  Interventions: Drug: Avenciguat (BI 685509)
- Placebo (Placebo Comparator): Participants in this dose group received matching placebo twice daily (BID) throughout the study period. At Visit 2 (Week 1), each dose consisted of one 1 mg placebo tablet and one 2 mg placebo tablet (four tablets daily). At Visit 3 (Week 2), a pseudo up-titration was implemented, maintaining the same tablets (one 1 mg and one 2 mg placebo per dose) for blinding. From Visit 4 onward (Week 3+), a second pseudo up-titration adjusted the dose to one 2 mg placebo tablet and one 3 mg placebo tablet per dose (four tablets daily). All doses were taken with water, with or without food.
  Interventions: Drug: Placebo matching Avenciguat (BI 685509)

INTERVENTIONS:
Drug: Avenciguat (BI 685509) — Participants received Avenciguat twice daily (BID) throughout the study. Up-titration depended on the assigned dose group. At Visit 2 (Week 1), each dose included one 1 mg Avenciguat tablet. At Visit 3 (Week 2), the dose was increased to one 2 mg Avenciguat tablet per dose. From Visit 4 onward (Week 3+), participants received one 3 mg Avenciguat tablet per dose. This regimen continued for 24 weeks, with all doses taken with water, with or without food.
  Arms: Avenciguat 2 mg BID; Avenciguat 3 mg BID
Drug: Placebo matching Avenciguat (BI 685509) — Participants received matching placebo twice daily (BID) throughout the study. At Visit 2 (Week 1), each dose included one 1 mg and one 2 mg placebo tablet (four tablets daily). A pseudo up-titration was applied at Visit 3 (Week 2), maintaining the same tablet composition to preserve blinding. From Visit 4 (Week 3) onward, a second pseudo up-titration adjusted each dose to one 2 mg and one 3 mg placebo tablet (four tablets daily). All doses were taken with water, with or without food.
  Arms: Placebo

SUMMARY:
This study is open to adults with liver cirrhosis and high blood pressure in the portal vein (main vessel going to the liver). The purpose of this study is to find out whether a medicine called Avenciguat helps people with this condition.

Participants are put into 3 groups randomly, which means by chance. Participants in 2 groups take different doses of Avenciguat as tablets twice a day. Participants in the placebo group take placebo as tablets twice a day. Placebo tablets look like Avenciguat tablets but do not contain any medicine.

Participants are in the study for about 8 months. During this time, they visit the study site about 14 times. At 3 of the visits, the doctors check the pressure in a liver vein. This is done with a catheter (a long thin tube) and gives information about the pressure in the portal vein. The change in blood pressure is then compared between the groups to see whether the treatment works.

The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
2. Male or female who is ≥ 18 (or who is of legal age in countries where that is greater than 18) and ≤ 75 years old at screening
3. Clinical signs of Clinically Significant Portal Hypertension (CSPH) as described by either one of the points below. Each trial patient must have a gastroscopy during the screening period or within 6 months prior to screening.

   * documented endoscopic proof of oesophageal varices and / or gastric varices at screening or within 6 months prior to screening
   * documented endoscopic-treated oesophageal varices as preventative treatment
4. CSPH defined as baseline Hepatic Venous Pressure Gradient (HVPG) ≥ 10 mmHg, based on a local interpretation of the pressure tracing
5. Diagnosis of compensated alcohol-related cirrhosis. Diagnosis must be based on histology (historical data is acceptable) or on clinical evidence of cirrhosis (e.g. platelet count < 150 x 10^9/L [150 x 10^3/µL], nodular liver surface on imaging or splenomegaly)
6. Abstinence from significant alcohol misuse / abuse for a minimum of 2 months prior to screening, and the ability to abstain from alcohol throughout the trial (both evaluated based on Investigator judgement)
7. Willing and able to undergo HVPG measurements per protocol (based on Investigator judgement)
8. If receiving statins must be on a stable dose for at least 3 months prior to screening, with no planned dose change throughout the trial Further inclusion criteria apply.

Exclusion Criteria:

1. Previous clinically significant decompensation events (e.g. ascites [more than perihepatic ascites], Variceal Haemorrhage (VH) and / or apparent Hepatic Encephalopathy (HE))
2. History of other forms of chronic liver disease (e.g. non-alcoholic steatohepatitis (NASH), Hepatitis B virus (HBV), untreated Hepatitis C Virus (HCV), autoimmune liver disease, primary biliary cholangitis, primary sclerosing cholangitis, Wilson's disease, haemachromatosis, alpha-1 antitrypsin (A1At) deficiency)
3. Has received curative anti-viral therapy with direct-acting anti-virals within the last 2 years for HCV, or, if such treatment was > 2 years ago and there is no sustained virological response (SVR) at screening, or, must take curative anti-viral therapy with direct-acting anti-virals throughout the trial
4. Alcohol-Related Liver Disease (ARLD) without adequate treatment (e.g. lifestyle modification) or with ongoing pathological drinking behaviour (misuse / abuse based on Investigator judgement)
5. Must take, or wishes to continue the intake of, restricted concomitant therapy or any concomitant therapy considered likely (based on Investigator judgement) to interfere with the safe conduct of the trial
6. Systolic Blood Pressure (SBP) < 100 mmHg and Diastolic Blood Pressure (DBP) < 70 mmHg at screening
7. Model of End-stage Liver Disease (MELD) score of > 15 at screening, calculated by the central laboratory
8. Hepatic impairment defined as a Child-Turcotte-Pugh score ≥ B8 at screening, calculated by the site, using central laboratory results Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (6):
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Floridian Clinical Research-Miami Lakes-68368, Miami Lakes, Florida
  - Northwell Health Center for Liver Disease, Manhasset, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
- Hospital Italiano de Buenos Aires, CABA, Argentina
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - AKH - Medical University of Vienna, Vienna
- Edegem - UNIV UZ Antwerpen, Edegem, Belgium
- Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec, Canada
- China (4):
  - Beijing Friendship Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - NanFang Hosptial, Guangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
- University Hospital Dubrava, Zagreb, Croatia
- Hvidovre Hospital, Hvidovre, Denmark
- France (2):
  - HOP d'Angers, Angers
  - HOP Rangueil, Toulouse
- Germany (3):
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
  - St. Josefs-Hospital, Wiesbaden, Wiesbaden
- Western Galilee Hospital, Nahariya, Israel
- Italy (4):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - Policlinico "Paolo Giaccone", Palermo
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Japan (5):
  - Shin-yurigaoka General Hospital, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Yokohama City University Hospital, Kanagawa, Yokohama
  - National Hospital Organization Yokohama Medical Center, Kanagawa, Yokohama
  - Osaka Metropolitan University Hospital, Osaka, Osaka
- Leids Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- ULS de Santa Maria, E.P.E, Lisbon, Portugal
- Regional Institute of Gastroenterology Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca, Romania
- Singapore General Hospital, Singapore, Singapore
- South Korea (2):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon State
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Puerta de Hierro, Majadahonda
- Ospedale Regionale di Lugano, Viganello, Switzerland
- Taipei Veterans General Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Once the time frame criteria given under number 4 are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Reiberger T, Berzigotti A, Trebicka J, Ertle J, Gashaw I, Swallow R, Tomisser A. The rationale and study design of two phase II trials examining the effects of BI 685,509, a soluble guanylyl cyclase activator, on clinically significant portal hypertension in patients with compensated cirrhosis. Trials. 2023 Apr 24;24(1):293. doi: 10.1186/s13063-023-07291-3. PMID 37095557
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind, placebo-controlled, parallel-group, multicenter trial included three treatment groups: two doses of avenciguat and a placebo, alongside standard care, in patients with clinically significant portal hypertension (CSPH) due to compensated alcohol-related cirrhosis. The primary objective was to estimate the mean difference in the percentage change in hepatic venous pressure gradient (HVPG) from baseline after 24 weeks. Safety and tolerability were also assessed.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Started (Randomized) | 26 | 27 | 27
Treated | 25 | 27 | 27
Completed (Completed trial medication) | 19 | 23 | 17
Not Completed | 7 | 4 | 10
Not completed — Withdrawal of consent | 0 | 1 | 1
Not completed — Study terminated by sponsor | 3 | 3 | 2
Not completed — Adverse Event | 3 | 0 | 6
Not completed — Randomised in error and was not treated | 1 | 0 | 0
Not completed — Subject decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomised set (RS) - this analysis set includes all enrolled patients that were randomised to the trial medication. One patient in the placebo group was randomised in error and was not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID | Total
Number analyzed (Participants) | 26 | 27 | 27 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (8.1) | 56.6 (9.2) | 57.1 (10.9) | 57.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 4 | 22
  Male | 17 | 18 | 23 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 3 | 16
  Not Hispanic or Latino | 22 | 18 | 24 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 21 | 21 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline hepatic venous pressure gradient (HVPG) [Mean (Standard Deviation); unit: Millimeter mercury (mmHg)] — Mean hepatic venous pressure gradient (HVPG) at baseline. Population: Full analysis set (FAS) - this analysis set includes all randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded.
  The one participant wrongly randomized in the placebo group was not included in this set.
  Millimeter mercury (mmHg)
    number analyzed (Participants) | 25 | 27 | 27 | 79
    (all) | 15.11 (4.10) | 14.95 (4.27) | 14.61 (4.07) | 14.88 (4.10)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Hepatic Venous Pressure Gradient (HVPG) From Baseline After 24 Weeks of Treatment
Description: HVPG was calculated as the difference between the average wedged hepatic venous pressure (WHVP) and either:
  Proximal Free Hepatic Venous Pressure (PFHVP), if judged more reliable, or Average Free Hepatic Venous Pressure (FHVP), if considered more reliable.
  Based on the central reader's judgment:
  If PFHVP was more reliable:
  HVPG(mmHg)= Average WHVP (mmHg) - PFHVP (mmHg)
  If FHVP was more reliable:
  HVPG(mmHg)=Average WHVP (mmHg)-Average FHVP (mmHg)
  Percentage Change = (HVPG at 24 weeks- Baseline HVPG/Baseline HVPG) × 100
  A restricted maximum likelihood (REML) approach using a mixed model with repeated measurements (MMRM) was used to estimate adjusted treatment means. The analysis included fixed categorical effects for treatment at each visit, use of non-selective beta-blockers (NSBBs) or carvedilol at baseline (yes/no), and fixed continuous effects for baseline hepatic venous pressure gradient (HVPG) at each visit.
Time Frame: From first administration of trial medication up to 24 weeks.
Population: Full analysis set (FAS) - this analysis set includes all randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded.
  The hypothetical strategy was used for handling intercurrent events for the primary objective as a main analysis as if all the intercurrent events had not happened.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Percentage of change | 7.07 [-6.07 to 20.21] | -1.33 [-13.41 to 10.75] | -7.11 [-22.02 to 7.80]
Statistical Analysis 1: Comparison: Placebo vs Avenciguat 2 mg BID; Model includes baseline HVPG as linear covariate and treatment and use of NSBBs or carvedilol as fixed effects, treatment by visit interaction and baseline HVPG by visit interaction. The following covariance structure has been used to fit the mixed model: Unstructured; Test type: Other — The adjusted mean values for percentage change at Week 24 are derived for each group using the MMRM. The mean difference for the "Comparison vs Placebo," is the adjusted mean of the treatment group subtracted from the adjusted mean of the placebo group; Difference of adjusted means = -8.40, 95% CI 2-sided [-26.25 to 9.45], Standard Error of Mean 8.90
Statistical Analysis 2: Comparison: Placebo vs Avenciguat 3 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Difference of adjusted means = -14.18, 95% CI 2-sided [-34.09 to 5.72], Standard Error of Mean 9.93

2. Secondary Outcome: Percentage Change in Hepatic Venous Pressure Gradient (HVPG) From Baseline, Measured in Millimeters of Mercury (mmHg), After 8 Weeks of Treatment
Description: HVPG was calculated as the difference between the average wedged hepatic venous pressure (WHVP) and either:
  Proximal Free Hepatic Venous Pressure (PFHVP), if judged more reliable. Average Free Hepatic Venous Pressure (FHVP), if considered more reliable.
  Based on the central reader's judgment:
  If PFHVP was more reliable:
  HVPG(mmHg)= Average WHVP (mmHg) - PFHVP (mmHg)
  If FHVP was more reliable:
  HVPG(mmHg)=Average WHVP (mmHg)-Average FHVP (mmHg)
  Percentage Change = (HVPG at 8 weeks- Baseline HVPG/Baseline HVPG) × 100
  This endpoint was analyzed using the Treatment Policy Estimand and an ANCOVA model. The model included baseline HVPG as a linear covariate, and treatment and use of non-selective beta-blockers (NSBBs) or carvedilol as fixed effects.
Time Frame: From first administration of trial medication up to 8 weeks.
Population: Full analysis set (FAS) - this analysis set includes all randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded.
  All intercurrent events (ICEs) were handled using the treatment policy for the secondary endpoints. That is, all data collected after the intercurrent events will be included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Percentage of change | -5.41 [-14.30 to 3.47] | -1.90 [-10.62 to 6.82] | -2.72 [-13.03 to 7.59]
Statistical Analysis 1: Comparison: Placebo vs Avenciguat 2 mg BID; The analysis of covariance (ANCOVA) model includes baseline hepatic venous pressure gradient (HVPG) as a linear covariate, with treatment and use of non-selective beta-blockers (NSBBs) or carvedilol as fixed effects. All intercurrent events (ICEs) will be handled using the treatment policy for the primary objective as a sensitivity analysis. That is, all data collected after the intercurrent events will be included in the analysis; Test type: Other — The adjusted mean values for percentage change at Week 8 are derived for each group using the MMRM. The mean difference for the "Comparison vs Placebo," is the adjusted mean of the treatment group subtracted from the adjusted mean of the placebo group; Difference of adjusted means = 3.51, 95% CI 2-sided [-8.94 to 15.96], Standard Error of Mean 6.23
Statistical Analysis 2: Comparison: Placebo vs Avenciguat 3 mg BID; ANCOVA) model includes baseline hepatic venous pressure gradient (HVPG) as a linear covariate, with treatment and use of non-selective beta-blockers (NSBBs) or carvedilol as fixed effects. All intercurrent events (ICEs) will be handled using the treatment policy for the primary objective as a sensitivity analysis. That is, all data collected after the intercurrent events will be included in the analysis; Test type: Other — [test comment as in outcome 2, analysis 1]; Difference of adjusted means = 2.69, 95% CI 2-sided [-10.94 to 16.33], Standard Error of Mean 6.82

3. Secondary Outcome: Response Defined as > 10% Reduction From Baseline HVPG (Measured in mmHg) After 8 Weeks of Treatment
Description: Response is defined as greater than 10% reduction from baseline HVPG (measured in mmHg) after 8 weeks of treatment. The number of participants with, or without response after 8 weeks of treatment with Avenciguat is reported.
Time Frame: From first administration of trial medication up to 8 weeks.
Population: Full analysis set (FAS) - this analysis set includes all randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded. If a patient misses the Week 8 visit, the missing data was not imputed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 24 | 25 | 18
Participants
  Yes | 10 | 10 | 7
  No | 14 | 15 | 11

4. Secondary Outcome: Response Defined as > 10% Reduction From Baseline HVPG (Measured in mmHg) After 24 Weeks of Treatment
Description: Response is defined as greater than 10% reduction from baseline HVPG (measured in mmHg) after 24 weeks of treatment.
Time Frame: From first administration of trial medication up to 24 weeks.
Population: Full analysis set (FAS) - this analysis set includes all randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded. If a patient misses the Week 24 visit, the missing data was not imputed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 19 | 23 | 17
Participants
  Yes | 5 | 11 | 4
  No | 14 | 12 | 13

5. Secondary Outcome: Occurrence of One or More Decompensation Events (i.e. Ascites, VH, and / or Overt HE) During the 24 Week Treatment Period
Description: A decompensation event is characterized by the occurrence of any of the following:
  * Ascites,
  * Variceal hemorrhage,
  * Overt hepatic encephalopathy.
Time Frame: From first administration of trial medication up to 24 weeks.
Population: Treated set (TS) - the treated set includes all patients who were randomised to the trial medication and were treated with at least one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Participants | 2 | 0 | 3

6. Secondary Outcome: Occurrence of CTCAE Grade 3 (or Higher) Hypotension or Syncope Based on Investigator Judgement, During the First 8 Weeks of the Treatment Period
Description: The occurrence of CTCAE grade 3 (or higher) hypotension or syncope, based on the investigator's judgment, during the first 8 weeks of the treatment period is reported.
Time Frame: From first administration of trial medication up to 8 weeks.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Participants | 0 | 0 | 1

7. Secondary Outcome: Occurrence of CTCAE Grade 3 (or Higher) Hypotension or Syncope Based on Investigator Judgement, During the 24 Week Treatment Period
Description: The occurrence of CTCAE grade 3 (or higher) hypotension or syncope, based on the investigator's judgment, during the 24 weeks of the treatment period is reported.
Time Frame: From first administration of trial medication up to 24 weeks.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Participants | 0 | 0 | 1

8. Secondary Outcome: Occurrence of Discontinuation Due to Hypotension or Syncope During the First 8 Weeks of the Treatment Period
Description: The occurrence of hypotension or syncope during the first 8 weeks of the treatment period leading to the participant's discontinuation is reported.
Time Frame: From first administration of trial medication up to 8 weeks.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Participants | 0 | 0 | 1

9. Secondary Outcome: Occurrence of Discontinuation Due to Hypotension or Syncope During the 24 Week Treatment Period
Description: The occurrence of hypotension or syncope during the first 24 weeks of the treatment period leading to the participant's discontinuation is reported.
Time Frame: From first administration of trial medication up to 24 weeks.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avenciguat 2 mg BID | Avenciguat 3 mg BID
Number analyzed (Participants) | 25 | 27 | 27
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: AE collection: From the first Avenciguat or placebo dose to the last dose, plus a 7-day residual effect period, totaling up to 182 days. All-cause mortality: From the first Avenciguat or placebo dose to the study's end, totaling up to 196 days.
Description: Treated set (TS) - the treated set includes all patients who were randomised to the trial medication and were treated with at least one dose.
Groups:
- Avenciguat 2mg BID: Participants received Avenciguat combined with matching placebo tablets twice daily (BID). At Visit 2 (Week 1), each dose included one 1 mg Avenciguat tablet and one 2 mg placebo tablet (four tablets daily). At Visit 3 (Week 2), the dose was up titrated to 2 mg Avenciguat BID (one 1 mg placebo tablet and one 2 mg Avenciguat tablet (four tablets daily)). From Visit 4 onward (Week 3+), a pseudo up-titration was applied, with participants taking one 2 mg Avenciguat tablet and one 3 mg placebo tablet per dose (four tablets daily) to maintain blinding. This regimen continued for 24 weeks, with doses taken with water, with or without food.
- Avenciguat 3mg BID: Participants received Avenciguat with matching placebo tablets twice daily (BID). At Visit 2 (Week 1), each dose contained one 1 mg Avenciguat tablet and one 2 mg placebo tablet (four tablets daily). At Visit 3 (Week 2), the dose was up titrated to 2 mg Avenciguat BID (one 1 mg placebo tablet and one 2 mg active tablet (four tablets daily)). From Visit 4 onward (Week 3+), the dose was further up titrated to 3 mg Avenciguat BID (one 2 mg placebo tablet and one 3 mg active tablet per dose (four tablets daily)). This regimen was maintained for 24 weeks, with doses taken with water, with or without food.
Arm/Group | Placebo | Avenciguat 2mg BID | Avenciguat 3mg BID
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/25 | 1/27 | 3/27
Other Adverse Events (participants affected / at risk) | 9/25 | 10/27 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Avenciguat 2mg BID (N=27) | Avenciguat 3mg BID (N=27)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Avenciguat 2mg BID (N=27) | Avenciguat 3mg BID (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 2 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 3
Headache (Nervous system disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 2
Hypotension (Vascular disorders) | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
This trial was discontinued after Boehringer Ingelheim ended Avenciguat's clinical development for CSPH due to lack of efficacy, not safety concerns. Enrollment was complete, but some patients were still in treatment. These patients were asked to stop trial medication and attend an Early Discontinuation Visit, then entered the follow-up period per the clinical trial protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05161481/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT05161481/SAP_001.pdf